CLINICAL TRIAL: NCT03077100
Title: Identification of Pathogens and Their Antibiogram in the Neonatal Intensive Care Unit (NICU)
Brief Title: Identification of Pathogens in the Neonatal Intensive Care Unit (NICU)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0001-17
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Pathogen Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborns with positive cultures: Positive cultures of newborns hospitalized in the NICU in the past 5 years will undergo laboratory examination and identification
  Interventions: Other: Laboratory identification of positive cultures

INTERVENTIONS:
Other: Laboratory identification of positive cultures — Laboratory identification of positive cultures

SUMMARY:
To aim of this study is to identify the pathogens and their distribution in the NICU and to determine whether empirical antibiotics are suitable for the treatment of sepsis in the unit.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with positive cultures

Exclusion Criteria:

-

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns hospitalized in NICU with positive cultures
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Antibiogram | One year
  Positive cultures will be examined using an antibiogram and pathogens will be identified

CONTACTS AND LOCATIONS:
Overall Officials: Michael Feldman, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No